CLINICAL TRIAL: NCT04396041
Title: Microvascular Plug (MVP) for the Treatment of Pulmonary ArterioVenous Malformations (PAVMs)
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00173822
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Arteriovenous Malformation
Keywords: Pulmonary Arteriovenous Malformation; PAVM; HHT; hereditary hemorrhagic telangiectasia
MeSH Terms: conditions — Pulmonary Arteriovenous Fistulas; Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients treated for Pulmonary Arteriovenous Malformation: All participants in the study will be patients who have been treated for Pulmonary Arteriovenous Malformation using Microvascular Plugs, Amplatzer Vascular Plugs or Detachable coils.
  Interventions: Device: Microvascular Plug (MVP); Device: Amplatzer Vascular Plug (AVP); Device: Detachable coils

INTERVENTIONS:
Device: Microvascular Plug (MVP) — Patient's Pulmonary AVM(s) treated via transcatheter embolization with Microvascular Plugs.
Device: Amplatzer Vascular Plug (AVP) — Patient's Pulmonary AVM(s) treated via transcatheter embolization with Amplatzer Vascular Plugs.
Device: Detachable coils — Patient's Pulmonary AVM(s) treated via transcatheter embolization with detachable coils.

SUMMARY:
The purpose of this study is to compare the use of the Micro Vascular Plug (MVP) system and other embolic devices in treatment of PAVMs. Pulmonary Arteriovenous Malformations (PAVMs) are abnormal connections between the pulmonary vein and the pulmonary artery. This affects blood flow between the heart and lungs which puts patients at risk of stroke, brain abscess, hypoxia and even sudden death. The standard treatment of PAVMs is embolization. Embolization is the placing of an embolic (synthetic agent) into a blood vessel to block blood flow. The embolic is inserted via a catheter into the blood vessel. Detachable coils are the most commonly used embolic in the treatment of PAVMs. Despite long procedure times, numerous coils that are often required to occlude a single PAVM and recanalization rates ranging from 5% to 15%, the most widely used embolic device is still the detachable coil.

DETAILED DESCRIPTION:
Transcatheter embolization has become the standard of care in the treatment of Pulmonary Arteriovenous Malformations (PAVMs). PAVM embolization is performed to prevent right to left shunting which puts patients at risk of stroke, brain abscess, hypoxia and even sudden death. Despite long procedure times, numerous coils that are often required to occlude a single PAVM and recanalization rates ranging from 5% to 15%, the most widely used embolic device is still the detachable coil delivered through a microcatheter. An alternative to coil embolization is the Amplatzer Vascular plug (AVP). AVPs allow for quick delivery of a single occluding device. AVPs, however, cannot be delivered through a microcatheter, limiting the AVPs' utility to larger PAVM with larger feeding arteries. The new MVPTM Micro Vascular Plug System (MVP, Medtronic) was designed to combine the best of both devices and allows for the occlusion of small vessels in a quick and predictable manner with a single embolic device through a micro catheter. At the investigators' institution the investigators have a very large PAVM practice, as the investigators are a large Hereditary Hemorrhagic Telangiectasia (HHT) center of excellence. Currently there is a paucity of data comparing these devices for the treatment of PAVMs. Specifically, there is little data to inform interventional radiologists' decision making process about which device to choose based on the patient's clinical characteristics, the size of the PAVM feeding artery, and cost.

The investigators will create a registry/database of all patients who undergo embolization for Pulmonary AVM at the investigators' HHT center of excellence collecting data and adding in data from the investigators' existing PAVM database dating back at least the last 7 years. Patients with MVP embolizations will be assessed and compared to patients who are embolized with other solid embolic devices (coils/plugs). The investigators will assess reperfusion rates, immediate technical success, procedural attributes including procedure time, fluoroscopy time, contrast administration, and finally embolic and overall procedural costs.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing embolization of Pulmonary Arteriovenous Malformation (PAVM)

Exclusion Criteria:

* PAVM unable to be embolized

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Pulmonary Arteriovenous Malformation (PAVM) being treated through the Interventional Radiology clinic.
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Reperfusion Rates | Up to 3 Years
  Analyzed at 1 year and 3 years. Based on the investigators' preliminary data, reperfusion has been seen at 1-2 years in the patients the investigators have treated with coils and AVP making the 3-year goal for the investigators' prospective analysis feasible to cover reperfusion.
Immediate post-procedural success | Immediately after procedure up to 5 minutes
  Immediate post-procedural technical success defined as complete occlusion of the feeding artery supplying the PAVM.

SECONDARY OUTCOMES:
Procedure duration | Up to 4 hours
  Duration of procedure in minutes.
Fluoroscopy time | Up to 4 hours
  Fluoroscopy time measured in minutes.
Contrast dose | Up to 4 hours
  Contrast dose in mL.
Cost of embolic device per PAVM | Up to 4 hours
  The number of embolic used per procedure will be used to determine the cost per PAVM.
Overall procedure cost for PAVM | Up to 1 week
  Overall procedure cost for PAVM will be determined at 1 week after the procedure.
Radiation Dose Area Product (DAP) | Up to 4 hours
  Radiation DAP measured in milligray-centimeters squared (mGy-cm^2).
Cumulative Air Kerma (AK) dose | Up to 4 hours
  Cumulative Air Kerma dose measured in milligray (mGy).

CONTACTS AND LOCATIONS:
Overall Officials: Clifford R Weiss, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States